CLINICAL TRIAL: NCT06282042
Title: Early Transcatheter Mitral Valve Repair After Myocardial Infarction
Acronym: EMCAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Principal Investigator, Isaac Pascual Calleja, MD, PhD, Fundación para la Investigación Biosanitaria del Principado de Asturias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMCAMI
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-12

CONDITIONS: Acute Mitral Regurgitation
Keywords: MitraClip

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, randomised, open-label, comparative effectiveness clinical trial for the treatment of clinically significant functional mitral regurgitation within 60 days after acute myocardial infarction, who are treated per standard of care and who have been determined by the site's local heart team as inappropriate or too high risk for mitral valve surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEER + OMT (Experimental): Early transcatheter edge-to-edge mitral valve repair (TEER) plus optimal medical treatment
  Interventions: Procedure: Early transcatheter edge-to-edge mitral valve repair (TEER).; Device: MitraClip; Other: Optimal medical treatment
- OMT (Other): Optimal medical treatment
  Interventions: Other: Optimal medical treatment

INTERVENTIONS:
Procedure: Early transcatheter edge-to-edge mitral valve repair (TEER). — TEER will be planned and performed as soon as possible, but within 60 days after index myocardial infarction, and within 30 days of randomisation using the MitraClip device.
  Arms: TEER + OMT
Device: MitraClip — MitraClip
  Arms: TEER + OMT
Other: Optimal medical treatment — Optimal medical treatment

SUMMARY:
To explore the impact of early transcatheter edge-to-edge repair of acute functional mitral regurgitation after myocardial infarction on the combined incidence of death and heart-failure associated hospitalisations at one-year follow-up, and quality of life and LV remodelling at two-year follow-up.

DETAILED DESCRIPTION:
Prospective, multicentre, randomised, open-label, comparative effectiveness clinical trial for the treatment of clinically significant functional mitral regurgitation within 60 days after acute myocardial infarction, who are treated per standard of care and who have been determined by the site's local heart team as inappropriate or too high risk for mitral valve surgery.

Eligible subjects will be randomized in a 1:1 ratio to the MitraClip device (intervention group) or to no MitraClip device (Control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic moderate to severe or severe MR after acute MI
* Age > 18 years
* Based on the following classification recently published in "Transcatheter Mitral Edge-to-Edge Repair for Treatment of Acute Mitral Regurgitation" by M. Shuvy et al. (Can J Cardiol. 2023) patients will be included if categorized in Type 2, 3 or 4:

Exclusion Criteria:

* Primary MR (e.g. papillary muscle rupture)
* EF ≤ 25%
* Accepted for CABG
* Presence of cardiogenic shock (AMR type 1)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2027-06-16 (Estimated); Study Completion 2028-06-16 (Estimated)

PRIMARY OUTCOMES:
All-cause death or Cumulative Heart Failure hospitalizations | 12 months
  Composite of
  1. All-cause death
  2. Cumulative Heart Failure hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Pascual, MD, PhD, Principal Investigator — Hospital Universitario Central de Asturias
Locations (32):
- Israel (4):
  - Emek Medical Center, Afula, Afula
  - Shaare Zedek Medical Center, Jerusalem, Jerusalen
  - Rabin Medical Center, Petah Tikva, Petah Tikva
  - Sheba Medical Center, Ramat Gan, Ramat Gan
- Italy (5):
  - Civil Hospital of Brescia, Brescia, Brescia
  - Ospedale Policlinico San Martino, Genova, Genova
  - San Raffaele Hospital, Milan, Milano
  - Centro Cardiológico Monzino, Milan, Milan
  - Policlínico San Donato, San Donato Milanese, San Donato Milanese
- Netherlands (8):
  - Amsterdam University Medical Center, Amsterdam, Amsterdam
  - Amphia Hospital, Breda, Breda
  - Catharina Ziekenhuis Hospital, Eindhoven, Eindhoven
  - Leiden University Medical Center, Leiden, Leiden
  - Maastricht University Medical Center, Maastricht, Maastricht
  - St. Antonius Hospital, Nieuwegein, Nieuwegein
  - Erasmus University Medical Center, Rotterdam, Rotterdam
  - Isala Hospital, Zwolle, Zwolle
- Spain (15):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Clínic Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Doctor Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pocock SJ, Ariti CA, Collier TJ, Wang D. The win ratio: a new approach to the analysis of composite endpoints in clinical trials based on clinical priorities. Eur Heart J. 2012 Jan;33(2):176-82. doi: 10.1093/eurheartj/ehr352. Epub 2011 Sep 6. PMID 21900289
- [Background] Finkelstein DM, Schoenfeld DA. Combining mortality and longitudinal measures in clinical trials. Stat Med. 1999 Jun 15;18(11):1341-54. doi: 10.1002/(sici)1097-0258(19990615)18:113.0.co;2-7. PMID 10399200
- [Background] Shuvy M, Maisano F, Strauss BH. Transcatheter Mitral Edge-to-Edge Repair for Treatment of Acute Mitral Regurgitation. Can J Cardiol. 2023 Oct;39(10):1382-1389. doi: 10.1016/j.cjca.2023.05.009. Epub 2023 May 18. PMID 37209883
- [Background] Shuvy M, von Bardeleben RS, Grasso C, Raake P, Lurz P, Zamorano JL, Asch F, Kar S, Maisano F; EXPAND Investigators. Safety and efficacy of MitraClip in acutely ill (NYHA Class IV) patients with mitral regurgitation: Results from the global EXPAND study. ESC Heart Fail. 2023 Apr;10(2):1122-1132. doi: 10.1002/ehf2.14273. Epub 2023 Jan 4. PMID 36599332
- [Background] Haberman D, Estevez-Loureiro R, Benito-Gonzalez T, Denti P, Arzamendi D, Adamo M, Freixa X, Nombela-Franco L, Villablanca P, Krivoshei L, Fam N, Spargias K, Czarnecki A, Pascual I, Praz F, Sudarsky D, Kerner A, Ninios V, Gennari M, Beeri R, Perl L, Wasserstrum Y, Danenberg H, Poles L, George J, Caneiro-Queija B, Scianna S, Moaraf I, Schiavi D, Scardino C, Corpataux N, Echarte-Morales J, Chrissoheris M, Fernandez-Peregrina E, Di Pasquale M, Regueiro A, Vergara-Uzcategui C, Iniguez-Romo A, Fernandez-Vazquez F, Dvir D, Maisano F, Taramasso M, Shuvy M. Conservative, surgical, and percutaneous treatment for mitral regurgitation shortly after acute myocardial infarction. Eur Heart J. 2022 Feb 12;43(7):641-650. doi: 10.1093/eurheartj/ehab496. PMID 34463727
- [Background] Jung RG, Simard T, Kovach C, Flint K, Don C, Di Santo P, Adamo M, Branca L, Valentini F, Benito-Gonzalez T, Fernandez-Vazquez F, Estevez-Loureiro R, Berardini A, Conti N, Rapezzi C, Biagini E, Parlow S, Shorr R, Levi A, Manovel A, Cardenal-Piris R, Diaz Fernandez J, Shuvy M, Haberman D, Sala A, Alkhouli MA, Marini C, Bargagna M, Schiavi D, Denti P, Markovic S, Buzzatti N, Chan V, Hynes M, Mesana T, Labinaz M, Pappalardo F, Taramasso M, Hibbert B. Transcatheter Mitral Valve Repair in Cardiogenic Shock and Mitral Regurgitation: A Patient-Level, Multicenter Analysis. JACC Cardiovasc Interv. 2021 Jan 11;14(1):1-11. doi: 10.1016/j.jcin.2020.08.037. Epub 2020 Oct 14. PMID 33069653